CLINICAL TRIAL: NCT07196787
Title: Prophylactic Exercise Therapy for Musculoskeletal Side Effects in Isotretinoin Users: A Controlled Study
Brief Title: Exercise Therapy for Isotretinoin Users
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Asli keles onal, MD, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Asli1
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Isotretinoin; Isotretinoin Adverse Reaction
Keywords: exercise; pain; prophylaxis; side effects
MeSH Terms: conditions — Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Controlled study
Who Masked: Outcomes Assessor
Masking Description: The physiotherapist performing the outcome measurements will be unaware of the study protocol and the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacroiliac (SI) joint exercise group (Experimental): This 18-week, 5-day-a-week program is a comprehensive plan designed to build stability, strength, and mobility progressively while being mindful of the sensitivity of the SI joint.
  This program is divided into three 6-week phases. Each week consists of 5 sessions, mixing different focuses to ensure balanced development.
  Day 1: Foundational Strength & Stability
  Day 2: Low-Impact Cardio & Active Recovery
  Day 3: Core Focus & Hip Stability
  Day 4: Low-Impact Cardio & Mobility
  Day 5: Full Body Integration & Strength
  Interventions: Other: Exercise
- Control group (No Intervention): Control group: No intervention

INTERVENTIONS:
Other: Exercise — The 18-Week Program Structure This program is divided into three 6-week phases. Each week consists of 5 sessions, mixing different focuses to ensure balanced development.
  Day 1: Foundational Strength & Stability
  Day 2: Low-Impact Cardio & Active Recovery
  Day 3: Core Focus & Hip Stability
  Day 4: Low-Impact Cardio & Mobility
  Day 5: Full Body Integration & Strength
  Arms: Sacroiliac (SI) joint exercise group

SUMMARY:
Isotretinoin (13-cis retinoic acid) is a retinoic acid that is a derivative of vitamin A. Isotretinoin has been used effectively alone in acne treatment for 35 years. However, it has many side effects. Among the musculoskeletal side effects of this treatment, acute sacroileitis is a common condition. In this clinical picture, recovery may last for a few months after discontinuation of isotretinoin treatment. However, it may become permanent in some cases. According to our current knowledge, there is no study in the literature that prescribes exercise therapy for this patient group. This study, planned to investigate the effects of stretching and sacroiliac mobilization exercises on musculoskeletal pain and quality of life, which are among the side effects of isotretinoin treatment.

DETAILED DESCRIPTION:
Isotretinoin (13-cis retinoic acid) is a vitamin A derivative of retinoic acid. It was approved by the FDA in 1982 for the treatment of severe, refractory nodulocystic acne. Isotretinoin has been used effectively alone in the treatment of acne for 35 years. Isotretinoin is used in a daily dose range of 0.5-1 mg/kg/day. Starting treatment with high doses increases the risk of acute exacerbation, inflammation and scarring and is not recommended. The side effects of this treatment are often dose-dependent and the most common side effects are related to the skin and mucous membranes. Hypervitaminosis A-related side effects affecting the skin, eye, neurologic, hepatic and skeletal-muscular system are available. On the skin; dryness, cheilitis, dryness in the eyes, epistaxis, itching, dryness in the eyes may be observed. Ocular findings include xerophthalmia, conjunctivitis, night blindness, keratitis and optic neuritis. Pseudotumor cerebri, a rare side effect, is characterized by severe headache, nausea and visual changes. As a result, side effects such as forgetfulness, headache, decreased concentration, menstrual irregularity, increased blood lipid and transaminase levels, myalgia, arthralgia and low back pain may be observed during isotretinoin use . Isotretinoin-associated bilateral or unilateral sacroiliitis is among other reported side effects. Sacroiliitis is usually seen as acute sacroiliitis days or weeks after the start of isotretinoin treatment. Recent literature suggests that the reduction of pro-inflammatory cytokines (e.g. TNF-α, IL-1β, IL-6) and the release of anti-inflammatory myokines (e.g. IL-6, IL-10) are the key mechanisms of exercise in inflammatory rheumatic diseases. In addition, the function of regulatory T-cells is enhanced by exercise, which also reduces oxidative stress and improves the function of these cells. A review of the benefits of exercise in PsA was carried out, with findings including reduced disease activity, improved physical function and decreased inflammation. Moreover, discourse is had on the psychological advantages of physical exertion, including a reduction in symptoms of depression and anxiety. The impact of exercise on AS was evaluated, with improvements in spinal mobility, pain and inflammation being emphasised. They also discuss the role of exercise. They discuss how exercise can reduce oxidative stress. They also discuss how exercise can improve cardiovascular health. They focus on this in relation to AS patients. So, the hypothesis of this study was predicated on the theory that regular exercise reduces disease burden by improving joint mobility, muscle strength and overall physical function, in addition to its salutary anti-inflammatory effects. The H1 hypothesis of this study was that regular exercise programmes have a favourable impact on the adverse musculoskeletal effects of isotretinoin treatment.

Material-Method:

In this study, it was planned to investigate the effects of stretching and sacroiliac mobilization exercises on musculoskeletal pain and sacroileitis, which are side effects of the drug, on musculoskeletal pain and quality of life in patients started on isotretinoin treatment. Between August 2025 and January 2026, patients who applied to the dermatology outpatient clinic and planned to start isotretinoin will be informed about the study, one group will be taught a sacroiliac stretching and mobilization exercise program and will be asked to perform these exercises 10 times in 2 sets every day. The other group will consist of patients who do not exercise and take medication. Within the scope of this prospectively planned study, it is planned to evaluate the patients by collecting data in 4 stages. The first stage will be collected before the start of isotretinoin treatment, the second stage in the 1st month of treatment, the third stage in the 3rd month of treatment and the last stage in the 6th month of treatment by evaluating pain measurement and quality of life. Musculoskeletal pain measurements, quality of life, and conditions occurring during follow-up will be evaluated and compared between the exercising group and the non-exercising group.

Pain measurement; The pain sensitivity of the subjects to pressure will be evaluated with a pain meter device called algometer. Algometer Commender Jtech Medical 801-478 USA brand digital algometer will be used in the evaluation. This device is already in current use and belongs to the researchers themselves. The algometer will be used to measure the trapezius muscle trunk, latissimus dorsi muscle trunk and sacroiliac joints bilaterally 3 times each. Before the measurement, the areas will be marked and the algometer will be placed perpendicular to these points and the subjects will be asked to report the first sensation of pain. The pain threshold will be recorded in pounds (1kg=2.2 pounds) by reading the value on the indicator.

Quality of Life measurement; World Health Organization Quality of Life (WHOQOL-SHORT FORM) is a statement-based measure developed to assess perception, personal goals, standards and concerns within one's own culture and values. The WHOQOL-SHORT FORM measures the following domains: physical health, psychological health, social relationships and environment. High scores indicate high quality of life, while low scores indicate low quality of life. Turkish validity and reliability has been realized (4).

Hypothesis(es): Regular exercises will have a positive effect on pain and quality of daily life levels in patients started on isotretinoin treatment.

ELIGIBILITY:
Inclusion Criteria:

* The participant is between the ages of 18-35,
* Not having a regular exercise habit,
* Starting Isotretinoin treatment for the first time.

Exclusion Criteria:

* Presence of any diagnosed rheumatologic disease,
* The presence of any diagnosed neurological disease,
* Having any diagnosed psychiatric illness,
* Having a physical disability that prevents them from exercising for any reason.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Pressure Algometer Testing | Baseline / first month / third month / sixth month
  Device: Jtech Medical 801/478 USA™ digital pressure algometer. Data collected and processed from the human algometer will generate a specific nociceptive response to neurostimulation in the somatosensory cortex.
  The algometer head was applied at a 90° angle to trigger points at selected locations, with pressure increased at a speed of approximately 100 g/s. One measurement was taken at the first sensation of pain, after which the process stopped.
Short Form 36 | Baseline / first month / third month / sixth month
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. Pricing depends on the number of scores that the researcher needs to calculate.

SECONDARY OUTCOMES:
VAS (visual analogue scale) | Baseline / first month / third month / sixth month
  The VAS is a unidimensional measure of pain intensity that is used to record patients' pain progression or to compare the severity of pain between patients with similar conditions. Numerical rating scales will be used. The score is determined by measuring the distance (in millimetres) on the 10-centimetre line between the 'no pain' anchor and the patient's mark. This provides a range of scores from 0 to 100. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Y Karahan, MD, Study Director — Uşak University
Locations (1):
- Usak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Research data supporting this publication are available upon request from the authors. The datasets generated and/or analyzed during the current study are available from the corresponding author; Ali Yavuz Karahan email: ali.karahan@usak.edu.tr / mobile: +905386921934.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From September 2026, the datasets created and/or examined during the present study will be accessible to the public from the person responsible for the study.
Access Criteria: Plan to Share IPD: "Yes" Plan Description: "No individual participant data will be shared. Results will be published by the investigators in academic journals.